CLINICAL TRIAL: NCT00514410
Title: Folate Augmentation of Treatment - Evaluation for Depression: a Randomised Controlled Trial
Acronym: FolATED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangor University (Other)
Collaborators: NHS Health Technology Assessment Programme (Other); Swansea University (Other); Cardiff University (Other); University of Liverpool (Other); North West Wales NHS Trust (Other); North East Wales NHS Trust (Other); Swansea NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G0373; ISRCTN37558856
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2009-02

CONDITIONS: Depression
Keywords: Depression; Folate; Folic acid; Antidepressants
MeSH Terms: conditions — Depression | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folic Acid (Experimental)
  Interventions: Drug: Folic Acid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folic Acid — Folic acid 5 mg once a day for three months as a supplement to their antidepressant treatment
  Arms: Folic Acid
Drug: Placebo — Matching placebo taken once a day for three months
  Arms: Placebo

SUMMARY:
To determine whether giving folic acid to people with depression will help their antidepressants work better. If folate does help antidepressants to work better, then it will provide a safe, simple and cheap way of improving the treatment of depression.

DETAILED DESCRIPTION:
Clinical depression is common, debilitating and treatable; one in four people experience it during their lives. The majority of sufferers are treated in primary care and only half respond well to active treatment. Evidence suggests that folate may be a useful adjunct to antidepressant treatment: 1) patients with depression often have a functional folate deficiency; 2) the severity of such deficiency, indicated by elevated homocysteine, correlates with depression severity, 3) low folate is associated with poor antidepressant response, and 4) folate is required for the synthesis of neurotransmitters implicated in the pathogenesis and treatment of depression.

The primary objective of this multi-centred placebo-controlled randomised trial is to estimate the effect of folate augmentation in new or continuing treatment of depressive disorder in primary and secondary care. Secondary objectives are to evaluate the cost-effectiveness of folate augmentation of antidepressant treatment, investigate how the response to antidepressant treatment depends on genetic polymorphisms relevant to folate metabolism and antidepressant response, and explore whether baseline folate status can predict response to antidepressant treatment.

Comparisons: Eligible patients with moderate to severe depression will be randomised to receive 5mg of folic acid or placebo as an adjunct to their antidepressant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Only patients aged 18 or over
* ICD-10 diagnosis of moderate to severe depression
* Able to give informed consent (not delirious, actively psychotic or with severe communication or learning disability)
* Able to complete the research assessments

Exclusion Criteria:

* are folate deficient
* are B12 deficient
* have knowingly taken supplements containing folic acid within 2 months
* suffer from psychosis
* are already participating in another research project
* are pregnant or planning to become pregnant
* are taking anticonvulsants
* have a serious, advanced or terminal illness with a life expectancy of less than 1 year
* have recently started treatment for a medical condition which has not yet been stabilised
* are taking lithium
* have had a diagnosis or treatment for any malignant disease or any related condition such as intestinal polyposis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Self rated symptoms of depression using the Beck Depression Inventory | Repeated measures up to 6 months after initiation of folic acid/placebo

SECONDARY OUTCOMES:
Clinician rated depression using the Montgomery-Asberg Depression Rating Scale | Repeated measures up to 6 months after initiation of folic acid/placebo
Clinician rated symptom severity using the Clinical Global Impression scale | Repeated measures up to 6 months after initiation of folic acid/placebo
Health status using the SF12 | Repeated measures up to 6 months after initiation of folic acid/placebo
Adverse events | Repeated measures up to 6 months after initiation of folic acid/placebo
Cost Utility using the EuroQol, resource use questionnaire and medication history | Repeated measures up to 6 months after initiation of folic acid/placebo
Folate status | Baseline, 3 months and 6 months
Homocysteine Status | Baseline, 3 months and 6 months
The interaction between any of the genetic polymorphisms in the folate pathway that predicts the severity of depression, response to antidepressants, and the response to folate supplementation | Baseline only
Compliance - using the number of tablets remaining at each follow up, dispensing records for folic acid or placebo, dates of repeat prescriptions, Morisky questionnaire, red cell folate and homocysteine levels | 12 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian T Russell, PhD, HonFRCGP, FRCP Edin, FFPH, Principal Investigator — Swansea University; Keith Lloyd, MBBS, MSc, MRC Psych, MSc, MD, Principal Investigator — Swansea University
Locations (3):
- United Kingdom (3):
  - North West Wales Trust, Bangor, Gwynedd
  - Swansea University, Swansea, Swansea
  - Cardiff University, Wrexham, Wrexham

REFERENCES:
- [Background] Roberts SH, Bedson E, Hughes D, Lloyd K, Menkes DB, Moat S, Pirmohamed M, Slegg G, Thome J, Tranter R, Whitaker R, Wilkinson C, Russell I. Folate augmentation of treatment - evaluation for depression (FolATED): protocol of a randomised controlled trial. BMC Psychiatry. 2007 Nov 15;7:65. doi: 10.1186/1471-244X-7-65. PMID 18005429